CLINICAL TRIAL: NCT04636749
Title: Erbium Vaginal Laser for the Treatment of Stress Urinary Incontinence - Randomized Single Blind Trial
Brief Title: Erbium Vaginal Laser for the Treatment of Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Naama Farago MD, MD, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0379-20-RMB-CTIL
Record Dates: First submitted 2020-11-10; First posted 2020-11-19 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erbium laser (Active Comparator): Treatment with Erbium laser
  Interventions: Device: Erbium laser
- Sham laser (Sham Comparator): Treatment with sham laser
  Interventions: Device: Sham laser

INTERVENTIONS:
Device: Erbium laser — Vaginal laser therapy
  Arms: Erbium laser
Device: Sham laser — Sham laser therapy
  Arms: Sham laser

SUMMARY:
Two arms of women who suffer from clinical stress urinary incontinence. Women will be divided randomly into two arms. One arm will be treated with vaginal Erbium laser and the second with Sham laser, three treatments each. Follow up will be done 6 and 12 months after the last treatment.

DETAILED DESCRIPTION:
Examine the efficacy of vaginal Erbium laser treatment for stress urinary incontinence (SUI) in compare to placebo.

Plenty of women suffer from SUI. It is a condition in which involuntary urine leakage occurs during exercise. This condition affects about 40% of all women and causes huge disturbance to daily life. There are plenty of risk factors, such as age, obesity and parity. We assume that the pathophysiology is related to hypermobility of the urethra due to damage to the surrounding tissue.

The treatment options vary from surgical interventional to conservative, each treatment has its own success rate and risk factors. An attempt to find effective treatment option has been made.

The use of laser for various gynecologic conditions are at rise. ERBIUM type laser works on the lamina propria layer and causes rejuvenation probably by strengthening collagen structures and creating new ones.

The efficacy and safety of vaginal laser therapy has been proven already, but in the field of SUI the numbers in each study were low and there was no control group.

In this study we desire to examine the effect of vaginal ERBIUM treatment on SUI in compare to placebo.

this is a randomized single blind control trial. 40 women will be included in the research group and 40 in the placebo group. Women will be assigned randomly to each group. They will be treated with vaginal laser probe, three treatments 4 weeks apart. Follow up visits will be performed 3, 6, and 12 months after the first treatment.

Effectiveness evaluation will be done by physical urodynamic examination before treatment and 6 month after finishing, by 24 hours pad test' cough test and by fulfilling questionnaires-

1. The Urogenital Distress inventory (UDI6)
2. The Female Sexual Function Index (FSFI)

ELIGIBILITY:
Inclusion Criteria:

women above 18 with SUI -

Exclusion Criteria:

1. Recurrent pelvic inflammatory disease
2. Vaginal operation in the previous year
3. Women with abnormal uterine bleeding
4. Women with diagnosed genital herpes infection
5. Any concurrent lower genital tract infection -

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-10-22 (Estimated); Study Completion 2022-10-22 (Estimated)

PRIMARY OUTCOMES:
Cough test | From enrollment up to 12 months post treatment
  Results of full bladder cough test
Pad test | From enrollment up to 12 months post treatment
  Results of 24 hour pad weighing test

SECONDARY OUTCOMES:
Urinary distress index 6 | From enrollment up to 12 months post treatment
  Results of Urinary distress index 6 questionnaire
Female sexual function | From enrollment up to 12 months post treatment
  Results of female sexual function index questionnaire
Urinary incontinence and sexuality | From enrollment up to 12 months post treatment
  Results of urinary incontinence and sexuality questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Naama Farago, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cervigni M, Gambacciani M. Female urinary stress incontinence. Climacteric. 2015;18 Suppl 1:30-6. doi: 10.3109/13697137.2015.1090859. PMID 26366798
- [Background] Padmanabhan P, Dmochowski R. Urinary incontinence in women: a comprehensive review of the pathophysiology, diagnosis and treatment. Minerva Ginecol. 2014 Oct;66(5):469-78. Epub 2014 Jul 31. PMID 25078140
- [Background] Itkonen Freitas AM, Rahkola-Soisalo P, Mikkola TS, Mentula M. Current treatments for female primary stress urinary incontinence. Climacteric. 2019 Jun;22(3):263-269. doi: 10.1080/13697137.2019.1568404. Epub 2019 Feb 18. PMID 30773062
- [Background] Kobashi KC, Albo ME, Dmochowski RR, Ginsberg DA, Goldman HB, Gomelsky A, Kraus SR, Sandhu JS, Shepler T, Treadwell JR, Vasavada S, Lemack GE. Surgical Treatment of Female Stress Urinary Incontinence: AUA/SUFU Guideline. J Urol. 2017 Oct;198(4):875-883. doi: 10.1016/j.juro.2017.06.061. Epub 2017 Jun 15. PMID 28625508
- [Background] Dwyer PL, Karmakar D. Surgical management of urinary stress incontinence - Where are we now? Best Pract Res Clin Obstet Gynaecol. 2019 Jan;54:31-40. doi: 10.1016/j.bpobgyn.2018.10.003. Epub 2018 Oct 30. PMID 30503362
- [Background] Saraswat L, Rehman H, Omar MI, Cody JD, Aluko P, Glazener CM. Traditional suburethral sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2020 Jan 28;1(1):CD001754. doi: 10.1002/14651858.CD001754.pub5. PMID 31990055
- [Background] Majaron B, Srinivas SM, Huang He, Nelson JS. Deep coagulation of dermal collagen with repetitive Er:YAG laser irradiation. Lasers Surg Med. 2000;26(2):215-22. doi: 10.1002/(sici)1096-9101(2000)26:23.0.co;2-o. PMID 10685095
- [Background] Greene D, Egbert BM, Utley DS, Koch RJ. In vivo model of histologic changes after treatment with the superpulsed CO(2) laser, erbium:YAG laser, and blended lasers: a 4- to 6-month prospective histologic and clinical study. Lasers Surg Med. 2000;27(4):362-72. doi: 10.1002/1096-9101(2000)27:43.0.co;2-h. PMID 11074514
- [Background] Vizintin Z, Lukac M, Kazic M, Tettamanti M. Erbium laser in gynecology. Climacteric. 2015;18 Suppl 1:4-8. doi: 10.3109/13697137.2015.1078668. PMID 26366793
- [Background] Okui N. Efficacy and safety of non-ablative vaginal erbium:YAG laser treatment as a novel surgical treatment for overactive bladder syndrome: comparison with anticholinergics and beta3-adrenoceptor agonists. World J Urol. 2019 Nov;37(11):2459-2466. doi: 10.1007/s00345-019-02644-7. Epub 2019 Jan 28. PMID 30687908
- [Background] Pergialiotis V, Prodromidou A, Perrea DN, Doumouchtsis SK. A systematic review on vaginal laser therapy for treating stress urinary incontinence: Do we have enough evidence? Int Urogynecol J. 2017 Oct;28(10):1445-1451. doi: 10.1007/s00192-017-3437-x. Epub 2017 Aug 2. PMID 28770296
- [Background] Shobeiri SA, Kerkhof MH, Minassian VA, Bazi T; IUGA Research and Development Committee. IUGA committee opinion: laser-based vaginal devices for treatment of stress urinary incontinence, genitourinary syndrome of menopause, and vaginal laxity. Int Urogynecol J. 2019 Mar;30(3):371-376. doi: 10.1007/s00192-018-3830-0. Epub 2018 Dec 6. PMID 30523374
- [Background] Fistonic I, Fistonic N. Baseline ICIQ-UI score, body mass index, age, average birth weight, and perineometry duration as promising predictors of the short-term efficacy of Er:YAG laser treatment in stress urinary incontinent women: A prospective cohort study. Lasers Surg Med. 2018 Jan 23. doi: 10.1002/lsm.22789. Online ahead of print. PMID 29360142
- [Background] Su CF, Chen GD, Tsai HJ. Preliminary outcome of non-ablative vaginal Erbium laser treatment for female stress and mixed urinary incontinence. Taiwan J Obstet Gynecol. 2019 Sep;58(5):610-613. doi: 10.1016/j.tjog.2019.07.006. PMID 31542080
- [Background] Ogrinc UB, Sencar S, Lenasi H. Novel minimally invasive laser treatment of urinary incontinence in women. Lasers Surg Med. 2015 Nov;47(9):689-97. doi: 10.1002/lsm.22416. Epub 2015 Sep 21. PMID 26388213
- [Background] Conte C, Jauffret T, Vieillefosse S, Hermieu JF, Deffieux X. Laser procedure for female urinary stress incontinence: A review of the literature. Prog Urol. 2017 Dec;27(17):1076-1083. doi: 10.1016/j.purol.2017.09.003. Epub 2017 Oct 21. PMID 29033365
- [Background] Lin KL, Chou SH, Long CY. Effect of Er:YAG Laser for Women with Stress Urinary Incontinence. Biomed Res Int. 2019 Jan 15;2019:7915813. doi: 10.1155/2019/7915813. eCollection 2019. PMID 30766886
- [Background] Gambacciani M, Torelli MG, Martella L, Bracco GL, Casagrande AG, Albertin E, Tabanelli S, Viglietta M, D'Ambrogio G, Garone G, Cervigni M. Rationale and design for the Vaginal Erbium Laser Academy Study (VELAS): an international multicenter observational study on genitourinary syndrome of menopause and stress urinary incontinence. Climacteric. 2015;18 Suppl 1:43-8. doi: 10.3109/13697137.2015.1071608. PMID 26366800
- [Background] Lin YH, Hsieh WC, Huang L, Liang CC. Effect of non-ablative laser treatment on overactive bladder symptoms, urinary incontinence and sexual function in women with urodynamic stress incontinence. Taiwan J Obstet Gynecol. 2017 Dec;56(6):815-820. doi: 10.1016/j.tjog.2017.10.020. PMID 29241926
- [Background] Lin HY, Tsai HW, Tsui KH, An YF, Lo CC, Lin ZH, Liou WS, Wang PH. The short-term outcome of laser in the management of female pelvic floor disorders: Focus on stress urine incontinence and sexual dysfunction. Taiwan J Obstet Gynecol. 2018 Dec;57(6):825-829. doi: 10.1016/j.tjog.2018.10.010. PMID 30545535